CLINICAL TRIAL: NCT06566209
Title: Positron Emission Tomography for the Detection of Subclinical Immune Checkpoint Inhibitor-Induced Myocarditis (PET-SIM): A Prospective, Single Center, Single Arm, Open Label Pilot Study
Brief Title: FDG-PET as an Imaging Modality to Diagnose and Risk Stratify Subclinical, Imaging Negative Ici-Myocarditis
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 24-001222; NCI-2024-06871 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Subclinical Immune Checkpoint Inhibitor-Induced Myocarditis; Myocarditis; ICI-Myocarditis; Solid Malignant Tumor; Hematologic Malignancy; Subclinical Myocarditis; Subclinical ICI-myocarditis
MeSH Terms: conditions — Myocarditis; Hematologic Neoplasms | interventions — Positron-Emission Tomography; Tomography, X-Ray Computed; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Experimental FDG PET/CT: Patients undergo 18F-FDG and 13N-ammonia PET/CT scan, blood sample collection and have their medical records reviewed on study.
  Interventions: Device: Fluorodeoxyglucose - Positron Emission Tomography (FDG-PET)

INTERVENTIONS:
Device: Fluorodeoxyglucose - Positron Emission Tomography (FDG-PET) — Receive 18F-FDG PET/CT
  Other Names: 18F-fluorodeoxyglucose positron emission tomography; Positron Emission Tomography; Computed Tomography; FDG-PET; Positron Emission Tomography-Computed Tomography (PET/CT)

SUMMARY:
The purpose of this pilot study is to evaluate Fluorodeoxyglucose - Positron Emission Tomography (FDG-PET) as an imaging modality to diagnose and risk stratify subclinical, imaging negative ICI-myocarditis, and to determine whether subclinical ICI-induced myocarditis is a distinct and clinically relevant entity with a risk of progression to fulminant myocarditis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of signing informed consent
* Any solid or hematologic malignancy undergoing treatment with ICI (either as a single agent or in combination with others)
* Ambulatory and able to complete a 48-72 hour high fat and low carbohydrate diet with 18 hours fasting (PET diet), 18F-FDG PET/CT scanning, as well as 13N-ammonia PET-CT myocardial perfusion imaging (part of the routine protocol of the investigation). These two studies will be done as part of the same imaging set.
* Willing to return to Mayo Clinic for ongoing follow-up
* Left ventricular ejection fraction (LVEF) ≥45%
* Cardiac MRI (CMR) without conclusive evidence of inflammation, coronary assessment available (either via cardiac computed tomography angiography, CCTA, or via coronary angiogram) Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial.

Exclusion Criteria:

* Fulminant myocarditis requiring steroid therapy
* CMR with definitive evidence of myocarditis
* Clinical presentation consistent with acute coronary syndrome (wall motion abnormalities consistent with a specific coronary distribution, coronary angiogram with a culprit lesion identified, patients requiring revascularization either with percutaneous coronary interventions or coronary artery bypass grafting).
* Patients unable to provide informed consent
* Patients unable to complete the diet preparation protocol
* Pregnancy (all women of child-bearing age and potential will have a negative pregnancy test within 48 hours of the PET/CT at screen and 6-month visit)
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male or female patients diagnosed with having a solid tumor or cancers in the blood and who are undergoing treatment with immune checkpoint inhibitors (ICI) either as a single agent or in combination with others.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Presennce of inflammation or scarring | Baseline; Up to 7 months
  Assessed by reviewing 18F-FDG PET/CT imaging for presence of inflammation, progression/regression of inflammation or scarring.

SECONDARY OUTCOMES:
Incidence of hospitalization | Up to 2 years
  Assessed by review of medical record for incidence of hospitalization
Cardiovascular Intensive Care Unit (CICU) Level of Care Days | Up to 2 years
  Assessed by reviewing medical record for number of days, if any, of CICU care.
Incidence of arrhythmias | Up to 2 years
  Assessed by reviewing medical record for incidence of cardiac arrhythmias.

CONTACTS AND LOCATIONS:
Overall Officials: Martin G. Rodriguez-Porcel, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials